CLINICAL TRIAL: NCT02692859
Title: A Randomized, Positive-controlled, Non-inferiority Phase III Clinical Trial of a Haemophilus Influenzae Type b (Hib) Conjugate Vaccine in Healthy Infants and Children
Brief Title: A Phase III Clinical Trial of a Haemophilus Influenzae Type b (Hib) Conjugate Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Collaborators: Chengdu Olymvax Biopharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PRO-201301
Record Dates: First submitted 2016-02-24; First posted 2016-02-26 (Estimated); Results first posted 2017-08-21 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-07

CONDITIONS: Haemophilus Influenza

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vaccine(Chengdu Olymvax Biopharmaceuticals Inc.) (Experimental): Hib conjugate vaccine
  Interventions: Biological: Hib conjugate vaccine
- Vaccine (Walvax Biotechnology Co., LTD.) (Active Comparator): Hib conjugate vaccine
  Interventions: Biological: Hib conjugate vaccine

INTERVENTIONS:
Biological: Hib conjugate vaccine — Children aged 3-5 months: 3-dose(0,28,56 d);Children aged 6-11 months: 2-dose(0,28 d);Children aged 1-5 years:one dose(0 d), 0.5ml for each dose

SUMMARY:
Haemophilus influenza type b (Hib) remains a serious global health threat associated with high mortality and morbidity in young children. In China, The overall impact of Hib-related infections and the extent of coverage of Hib conjugate vaccines are unclear.Generally, vaccination has been considered the most effective way to prevent infection against Hib.In order to evaluate safety and immunogenicity of a haemophilus influenzae type b (Hib) conjugate vaccine developped by Chengdu Olymvax Biopharmaceuticals Inc. a phase III clinical trial is planned to conduct in healthy infants and children in China.

DETAILED DESCRIPTION:
Haemophilus influenza type b (Hib) remains a serious global health threat associated with high mortality and morbidity in young children. In China, The overall impact of Hib-related infections and the extent of coverage of Hib conjugate vaccines are unclear.Generally, vaccination has been considered the most effective way to prevent infection against Hib.In order to evaluate safety and immunogenicity of a haemophilus influenzae type b (Hib) conjugate vaccine developped by Chengdu Olymvax Biopharmaceuticals Inc. a randomized, positive-controlled, non-inferiority phase III clinical trial is planned to conduct in healthy infants and children in China.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 3-5 months/ 6-11 months/ 1-5 y for each age group
* Without vaccination history of Hib conjugate vaccine
* One of his/her guardians is able to understand and sign the informed consent
* Subjects' guardian can and will comply with the requirements of the protocol
* Subjects with temperature <=37.0°C on axillary setting

Exclusion Criteria:

* Subject who has a medical or family history of any of the following: allergic history, seizure, epilepsy, brain or mental disease
* Subject who is allergic to any ingredient of the vaccines
* Subject with damaged or low immune function which has already been known
* Subject who had a Hib disease medical history
* Subject with acute febrile illness or infectious disease
* Major congenital defects, developmental disorders or serious chronic illness
* Thrombocytopenia, blood coagulation disorder or bleeding difficulties with intramuscular injection
* Subject who has serious allergic history
* Subject with other medical history not suitable for vaccination such as difficulty for blood collection
* Any prior administration of immunodepressant or corticosteroids in last 6 months
* Any prior administration of blood products in last 3 months
* Any prior administration of other research medicine/vaccine in last 30 days
* Any prior administration of any attenuated live vaccine in last 14 days
* Any prior administration of subunit or inactivated vaccines in last 7 days, such as pneumococcal vaccine
* Any medical, psychological, social or other condition judged by investigator, that may interfere subject's compliance with the protocol or his/her guardian's signature on informed consent

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1992 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaccine(Chengdu Olymvax Biopharmaceuticals Inc.); Vaccine (Walvax Biotechnology Co., LTD.): Hib conjugate vaccine
  Hib conjugate vaccine: Children aged 3-5 months: 3-dose(0,28,56 d);Children aged 6-11 months: 2-dose(0,28 d);Children aged 1-5 y:one dose(0 d), 0.5ml for each dose
Period: Overall Study
Arm/Group | Vaccine(Chengdu Olymvax Biopharmaceuticals Inc.) | Vaccine (Walvax Biotechnology Co., LTD.)
Started | 996 | 996
Completed | 912 | 901
Not Completed | 84 | 95

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccine(Chengdu Olymvax Biopharmaceuticals Inc.) | Vaccine (Walvax Biotechnology Co., LTD.) | Total
Number analyzed (Participants) | 996 | 996 | 1992
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 996 | 996 | 1992
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months]
  12-60 months | 38.52 (12.84) | 37.32 (13.92) | 37.92 (13.44)
  6-11 months | 8.31 (1.80) | 8.20 (1.80) | 8.26 (1.80)
  3-5 months | 4.26 (0.82) | 4.27 (0.83) | 4.27 (0.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 481 | 464 | 945
  Male | 515 | 532 | 1047
Region of Enrollment [Number; unit: participants]
  China | 996 | 996 | 1992

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Adverse Reactions
Description: Number of Participants with Solicited Adverse Reactions
Time Frame: 0-7 days after each dose
Population: A total of participants in aged 3-5 months,6-11months and 1-5years
Measure: Number; unit: Count of Participants
Arm/Group | Vaccine(Chengdu Olymvax Biopharmaceuticals Inc.) | Vaccine (Walvax Biotechnology Co., LTD.)
Number analyzed (Participants) | 996 | 996
Count of Participants | 507 | 480

2. Primary Outcome: Proportion of Vaccinees With Anti-polyribosylribitol Phosphate (PRP) Concentrations ≥1.0μg/ml
Time Frame: 28 days after full course of vaccination
Reporting Status: Not Posted, anticipated posting 2017-12

3. Secondary Outcome: Incidence of Unsolicited Adverse Reactions
Time Frame: 0-28 days after each dose
Reporting Status: Not Posted

4. Secondary Outcome: Incidence of Serious Adverse Event (SAE) During the Whole Study Period
Time Frame: 0-84 days for children aged 3-5 months, 0-56 days for children aged 6-11 months and 0-28 days for children aged 1-5 y
Reporting Status: Not Posted

5. Secondary Outcome: Proportion of Vaccinees With Anti-polyribosylribitol Phosphate (PRP) Concentrations ≥0.15μg/ml
Time Frame: 28 days after full course of vaccination
Reporting Status: Not Posted

6. Secondary Outcome: the Anti-PRP Geometric Mean Concentrations (GMCs)
Time Frame: 28 days after full course of vaccination
Reporting Status: Not Posted

7. Secondary Outcome: the Anti-PRP Geometric Mean Fold Increase (GMFI)
Time Frame: 28 days after full course of vaccination
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Vaccine(Chengdu Olymvax Biopharmaceuticals Inc.) | Vaccine (Walvax Biotechnology Co., LTD.)
Serious Adverse Events (participants affected / at risk) | 10/996 | 15/996
Other Adverse Events (participants affected / at risk) | 0/996 | 0/996
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine(Chengdu Olymvax Biopharmaceuticals Inc.) (N=996) | Vaccine (Walvax Biotechnology Co., LTD.) (N=996)
bronchopneumonia (Infections and infestations) | 6 (6) | 12 (12)
upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
hand-foot-and-mouth disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
pneumonia (Infections and infestations) | 1 (1) | 1 (1)
viral enteritis (Gastrointestinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No